CLINICAL TRIAL: NCT07320677
Title: Finding Heart Failure in Those Prescribed Loop Diuretics in Primary Care in Jersey (FIND-HF LOOP)
Brief Title: Finding Heart Failure in Those Prescribed Loop Diuretics in Primary Care in Jersey
Acronym: FIND HF LOOP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Government of Jersey (Other Government)
Responsible Party: Principal Investigator, Aaron Henry, Cardiology Research Fellow, Government of Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025HCJREC03
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Diuretics
Keywords: NT-proBNP; Natriuretic peptide; Heart Failure; Screening
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - NTproBNP Screening (Experimental): Half of the island's GP surgeries will be randomly allocated to the intervention arm, whereby patients receiving a loop diuretic but without a diagnosis of heart failure or natriuretic peptide testing will be invited for a point of care NT-proBNP test.
  Interventions: Diagnostic Test: NT-proBNP screening
- Control - Usual care (No Intervention): Half of the island's GP surgeries will be randomly allocated to the control arm, whereby patients will continue with usual clinical care and won't be approached by the study team.

INTERVENTIONS:
Diagnostic Test: NT-proBNP screening — Patients in the intervention arm will be invited for a free point of care NT-proBNP blood test
  Arms: Intervention - NTproBNP Screening

SUMMARY:
The goal of this clinical trial is to learn whether a simple blood test screening pathway can help diagnose heart failure earlier in adults in primary care who take loop diuretic medicines (such as furosemide or bumetanide) but do not have a recorded diagnosis of heart failure.

The main questions it aims to answer are:

1. Does offering a NT-proBNP blood test to eligible patients increase the number of new heart failure diagnoses within 12 months compared with usual care?
2. Does this screening pathway also uncover other important heart problems, such as irregular heart rhythms (arrhythmias) or valve disease?

This is a cluster randomised controlled trial, which means that whole GP practices, rather than individual patients, are randomly assigned to one of two approaches:

1. NT-proBNP screening pathway, in which eligible patients are invited for a NT-proBNP blood test
2. Usual care, in which patients continue to be managed as they normally would without proactive screening

Participants will:

Be identified from GP records if they are prescribed loop diuretics and have no prior diagnosis of heart failure

In screening practices, be invited to attend for a free finger-prick NT-proBNP blood test and brief questionnaire

Be referred to the heart failure team and invited for an echocardiogram (a heart ultrasound scan) and further assessment if their NT-proBNP level is higher than 125 pg/mL

Researchers will compare outcomes between screening and usual-care practices after 12 months, focusing on new diagnoses of heart failure. They will also look at other important cardiovascular findings, such as new arrhythmias, valve disease, and heart failure hospitalisation rates.

ELIGIBILITY:
Inclusion Criteria:

* Receiving a loop diuretic (furosemide, bumetanide or torsemide)
* No coded diagnosis of heart failure in GP records
* Never had a natriuretic peptide test
* Willing to have a blood test for NT-proBNP

Exclusion Criteria:

* Clinical Frailty Score 7 or above on Rockwood frailty scale
* Prior diagnosis of heart failure
* Prior natriuretic peptide testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
New Heart Failure diagnosis at 12 months | 12 months from practice enrollment

SECONDARY OUTCOMES:
New clinically relevant cardiovascular disease | 12 months
  This will include moderate valvular disease and arrhythmia (eg, AF).
Heart Failure Hospitalisations | 12 months
All cause mortality | 12 months

OTHER OUTCOMES:
Number of patients with heart failure but not coded in primary care record | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jersey General Hospital, Saint Helier, Jersey